CLINICAL TRIAL: NCT05227495
Title: Effects of the Fully Immersive Leisure-based Virtual Reality Cognitive Training for Community-dwelling Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202100553B0
Record Dates: First submitted 2022-01-23; First posted 2022-02-07 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-01

CONDITIONS: Community-dwelling Elderly; Virtual Reality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental)
  Interventions: Behavioral: VR cognitive training
- control group (Active Comparator)
  Interventions: Behavioral: Traditional cognitive training

INTERVENTIONS:
Behavioral: VR cognitive training — All participants will receive trainings for 60 minutes per day, two days per week for 16 sessions.
  They will receive one immersive leisure-based VR cognitive training for 40 minutes. VR cognitive training receives four gardening activities.
  The cognitive elements including attention, working memory, processing speed, and executive function incorporated training.
  Arms: VR group
Behavioral: Traditional cognitive training — All participants will receive trainings for 60 minutes per day, two days per week for 16 sessions.
  The control group is performing traditional cognitive training program.
  Arms: control group

SUMMARY:
This study aims to (1) determine the feasibility and usability of immersive leisure-based VR cognitive training; (2) identify the intervention effects of immersive leisure-based VR cognitive training on cognitive function, daily function, and quality of life for elderly with community-dwelling elderly

DETAILED DESCRIPTION:
Cognitive training integrated into leisure activities can increase the training motivation of the elderly, while improving cognitive performance and daily functions. Virtual reality (VR) can simulate daily living situations, and it can be an effective intervention with cognitive training. Although a few studies have found immersive VR cognitive training can improve the cognitive function of the elderly with cognitive decline, these studies have shown inconsistent results. In addition, it is yet not clear the long-term effect of fully immersive VR cognitive training and its impact on daily function. Furthermore, for immersive VR cognitive training, there is still a lack of training programs that integrate into the context of leisure activities. This type of VR cognitive training could help the effectiveness of cognitive training to be transferred into daily functions.

ELIGIBILITY:
Inclusion Criteria:

1. age>=60
2. able to follow instruction
3. MMSE>=21

Exclusion Criteria:

1. dizziness or epilepsy history;
2. neurological or other orthopedic diseases with neurological or other orthopedic diseases (3)unstable physical condition of VR cognitive training;

(4)Recent psychiatric diagnosis, such as depression

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change scores of the Montreal Cognitive Assessment (MoCA) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Change scores of Wechsler Memory Scale (WMS) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  Including Faces Recognition (total scale=48), Verbal Paired Associates (total scale = 32), Word Lists (total scale = 48), Memory Span (total scale=48),and Spatial Span (total scale=32) will be used to assess the immediate, delayed, and working memory tests. For each subtest, a higher number indicates better performance in memory function. The raw score of subtests will also be transferred to standardized Z scores and summed to represent an index of general memory function.
Change scores of Stroop test | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. The time to complete the task will be calculated for each condition
Change scores of Color trials test | baseline, after the intervention eight weeks, and at 3-month follow-up.
  For Part 1, the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2, the respondent rapidly connects numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.

SECONDARY OUTCOMES:
Change scores of Wechsler Adult Intelligence Scale; WAIS | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The dual-task tests will be assessed to determine the ability for an individual to perform 2 tasks simultaneously. The investigators will assess the dual-task performance during walking and performing box and block test. The results of the dual-task tests will provide information regarding to whether the 2 tasks compete for the same class of neural resources or one of the tasks can be carried out automatically
Change scores of Everyday Cognition scales (ECog)-12 items | baseline, after the intervention eight weeks, and at 3-month follow-up.
  To detect cognitive and functional decline. The ECog shows promise as a useful tool for the measurement of general and domain-specific everyday functions in the elderly. There are six domains (Everyday Memory, Language, Visuospatial Abilities, Planning, Organization, and Divided Attention) in ECog. Lower scores represent a higher level of function in daily life.
Change scores of Amsterdam Instrumental Activity of Daily Living,A-IADL | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Amsterdam Instrumental Activity of Daily Living (A-IADL) is an adaptive and computerized questionnaire designed to assess impairments in instrumental activities of daily living (IADL) in (early) dementia. The questionnaire is completed by a caregiver, such as a relative or friend.
  Each item has a 5-point scale response option (scored 0-4). The scoring of the Amsterdam Instrumental Activity of Daily Living is calculated using item response theory .Lower scores indicating poorer performance.
Change scores of the World Health Organization Quality of Life-Old(WHOQOL-OLD) Taiwan Version | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The World Health Organization Quality of Life-Old questionnaires demonstrate acceptable psychometric performance in a convenience sample of Taiwan older people. It are valuable measures of Quality of Life-Old for use with older people.Time frame for assessment is the past two weeks.
  The items are distributed into 4 domains (physical; psychological, social and environmental health) and 25 facets.
Change scores of Community Integration Questionnaire, CIQ | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The community integration questionnaire (CIQ) was designed to assess home integration, social integration and productive activity in persons with acquired brain injury. The instrument consists of 15 items and can be completed by self report or with the assistance of a family member or caregiver familiar with the person's health status and social activities.
Change scores of Geriatric Depression Scale (GDS) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Geriatric Depression Scale (GDS) - 15 items version is a self-administered questionnaire used to evaluate mood and depressive symptoms. The scores range is 0-15 and a score of 5 or greater taken as a possible indicator of depression.
Change scores of The Chinese Aging Well Profile (CAWP) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  It comprised eight open-ended questions focusing on the meaning and interpretation of 'subjective well-being', e.g., 'Can you tell me what the important contributors to your well-being are?', 'Can you describe the important elements in your life that make you feel happy?', 'Can you describe the important elements in your life that you dislike?' and 'What does well-being personally mean to you?' To adapt the Aging Well Profile for a Chinese population in Taiwan was secured. It was agreed that the new version would be called the Chinese Aging Well Profile (CAWP).
Change scores of The Clinical Frailty Scale (CFS) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill). The aim of this scoping review is to identify and document the nature and extent of research evidence related to the CFS.
Change scores of Timed up and go (TUG) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The TUG assesses the dynamic balance ability and mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers in frail elderly (Podsiadlo & Richardson, 1991). The test-retest reliability of TUG on individuals with cognitive impairment was excellent (Blankevoort, van Heuvelen, & Scherder, 2013).
Change scores of 30 second chair stand test,CST | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The 30 second sit-to-stand will be assessed to indicate the strength and endurance level of the lower extremities. The 30 second sit-to-stand was standardized to allow hand support during the rise to and descent from standing but required participants to let go of the armrests with each stand. The participants will be asked to stand up from a standardized chair and then sit down as many times as possible within 30 seconds. The feasibility and reliability of using sit-to-stand test in people with cognitive impairment have been established to be good.
Change scores of Grip strength | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The investigator will use hand dynamometer to measure grip strength of both hands while the participant is seated, with the elbow at 90-degree flexion. The investigator will record the mean value of 3 attempts.
  Grip strength was measured using a digital dynamometers method, which is a tool with an adjustable grip span, ranging from 3.5 to 7 cm and weighing from 5 to 100 kg with minimal difference around 0.1 kg . All the participants were in a sitting position with fully extended elbows . Then, the investigator measured Grip strength on the dominant hand after 2-3 minutes of resting.
Change scores of short physical performance battery,SPPB | baseline, after the intervention eight weeks, and at 3-month follow-up.
  The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons. The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests . It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Change scores of Reported Edmonton Frail Scale (REFS) | baseline, after the intervention eight weeks, and at 3-month follow-up.
  Reported Edmonton Frail Scale is an adaptation of Edmonton Frail Scale, that can be performed in less than 10 min by any healthcare professional. Reported Edmonton Frail Scale substitutes the last domain on Edmonton Frail Scale, the physical performance measure, with three self-assessed physical performance questions . This is ideal for use in busy cardiology clinics when patients are being assessed for suitability for intervention. Scoring for the Reported Edmonton Frail Scale range is 0 to18. Not Frail：0-5 ;Apparently Vulnerable：6-7; Mildly Frail：8-9;Moderate Frailty：10-11;Sever Frailty：12-18.
Change scores of WHOQOL-bref Taiwan Version | baseline, after the intervention eight weeks, and at 3-month follow-up.
  As with the standard WHOQOL-BREF questionnaires the WHOQOL-BREF Taiwan version was simplified from the WHOQOL long form for Taiwan. For the purpose of cross-cultural comparison, the first 26 items were the same as the standard WHOQOL-BREF, which was developed from global studies. In addition to the 26 items, we applied the psychometric criteria proposed by the WHOQOL Group to select two more items from each of the two new facets to form the WHOQOL-BREF Taiwan version using data from the same 1,068 subjects. The selection process used for national items is described in the Results section. Thus, the WHOQOL-BREF Taiwan version contains 28 items classified into the same four domains as the standard WHOQOL-BREF. The scale administration and scoring procedures are the same as for the WHOQOL long form except that the facet score is based on only one item.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan